CLINICAL TRIAL: NCT03379844
Title: Holmium-166-radioembolization in Patients With Unresectable Hepatocellular Carcinoma (HCC); a Multi-center, Interventional, Non-randomized, Non-comparative, Open Label, Early Phase II Study: HEPAR Primary
Brief Title: HEPAR Primary: Holmium-166-radioembolization in Hepatocellular Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Cancer Society (Other); Erasmus Medical Center (Other); Quirem Medical B.V. (Industry)
Responsible Party: Principal Investigator, Marnix Lam, Prof, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL52338.041.17
Record Dates: First submitted 2017-11-21; First posted 2017-12-20 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Carcinoma Non-resectable
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Holmium-166 radioembolization (Experimental)
  Interventions: Device: Holmium-166 radioembolization

INTERVENTIONS:
Device: Holmium-166 radioembolization — An intra-arterial radioembolization procedure will be performed. The hepatic artery catheter is inserted via the femoral or radial artery under x-ray guidance by a trained interventional radiologist. The radiologist must repeatedly check the position of the catheter during the procedure to ensure it remains correctly sited and that reflux of the QuiremSpheres® into other organs does not occur. This is performed by injecting contrast medium. At the conclusion of the procedure, the catheter is removed.

SUMMARY:
Patients with hepatocellular carcinoma often die from intrahepatic disease since current treatment options are generally limited. Local treatment using holmium radioembolization could offer an effective treatment and a more personal approach than yttrium radioembolization (standard-of-care) as holmium has more imaging options.

DETAILED DESCRIPTION:
Primary objective:

• To establish the safety and toxicity profile of holmium radioembolization in patients with hepatocellular carcinoma.

Secondary objectives:

* To evaluate efficacy of holmium radioembolization in hepatocellular carcinoma without curative treatment options in a non-comparative phase II study.
* To evaluate tumor marker response.
* To evaluate Quality of Life (QoL).
* To evaluate biodistribution / dosimetry.
* To evaluate hepatic function.

Study design: Multi-center, interventional, treatment, non-randomized, open label, non-comparative, early phase II study. The study is a collaboration between UMC Utrecht and Erasmus MC Rotterdam. Recruitment and treatment of patients will take place in both centers.

Intervention: Holmium radioembolization will be performed via a catheter during angiography.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given written informed consent.
* Female or male aged 18 years and over.
* Diagnosis of HCC established according to the Netherlands HCC guideline criteria (in line with American AASLD criteria): nodule >1 cm in a patient at risk for HCC, with combination of arterial hypervascularity and venous or delayed phase wash-out on multiphase CT-scan or MRI-scan.2, 4 LR-5 and LR- 4 based on Liver Imaging Reporting and Data System can be included based on discretion of the principal investigator.I
* No curative treatment options (resection, transplant, or in case of solitary tumor <5 cm, RFA).
* Life expectancy of at least 6 months.
* ECOG Performance status 0-1 (Table 2).
* Liver-dominant disease (maximum 5 lung nodules all ≤1.0 cm and mesenteric or portal lymph nodes all ≤2.0 cm are accepted).
* Child-Pugh class A5-6 or B7.
* At least one measurable liver lesion according to the modified RECIST criteria.21
* Negative pregnancy test for women of childbearing potential. Female patients of child-bearing potential should use an highly effective acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) or should be more than 1 year postmenopausal or surgically sterile during their participation in this study (from the time they sign the consent form), to prevent pregnancy.

Exclusion Criteria:

* Evidence of significant extrahepatic disease (MRI-scan liver and multiphase abdominal CT as well as a thoracic CT are routinely performed at screening).
* Radiation therapy within the last 4 weeks before the start of study therapy.
* Previous or current treatment with RE. Previous treatment with TACE, surgery, RFA, and previous or current treatment with sorafenib are allowed.
* Major surgery within 4 weeks or incompletely healed surgical incision before starting study therapy.
* Serum bilirubin >34.2 micromole/L (2 mg/dL).
* Glomerular filtration rate <35 ml/min, determined according to the Modification of Diet in Renal Disease formula.
* Non-correctable INR >1.5 in case of femoral approach (as opposed to radial).
* Leukocytes <2 109/l and/or platelet count <50 109/l.
* Significant cardiac event (e.g. myocardial infarction, superior vena cava (SVC) syndrome, New York Heart Association (NYHA) classification of heart disease ≥2 within 3 months before entry, or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* Pregnancy or breastfeeding.
* Patients suffering from psychic disorders that make a comprehensive judgment impossible, such as psychosis, hallucinations and/or depression.
* Patients who are declared incapacitated.
* Previous enrollment in the present study.
* Male patients who are not surgically sterile or do not use an acceptable method of contraception during their participation in this study (from the time they sign the consent form) to prevent pregnancy in a partner.
* Evidence of untreated, clinically significant grade 3 portal hypertension (i.e. large varices at oesophago-gastro-duodenoscopy). In these cases, therapy with non-selective beta blocker (propranolol) or rubber band ligation should be instituted according to accepted guidelines. In case of small varices, prophylactic propranolol is advised.
* Portal vein thrombosis (tumor and/or bland) of the main branch (diagnosed on contrast enhanced transaxial images). Involvement of the right or left portal vein branches and more distal is accepted.
* Untreated active hepatitis. In case of detectable viral HBV load, treatment with a nucleos(t)ide analog such as entecavir or tenofovir should be instituted.
* Transjugular intrahepatic portosystemic shunt (TIPS).
* Body weight over 150 kg (because of maximum table load).
* Severe allergy for intravenous contrast used (Visipaque®)(because of CT evaluation, pre-treatment angiography and treatment angiography).
* Lung shunt >30 Gy, as calculated using scout dose SPECT/CT.
* Uncorrectable extrahepatic deposition of scout dose activity. Activity in the falciform ligament, portal lymph nodes and gallbladder is accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Safety, expressed as the rate of unacceptable toxicity. | Up to 6 months
  Safety, expressed as the rate of unacceptable toxicity, which is the occurrence of RE-induced liver disease, defined as a total bilirubin increase grade 3 or higher according to the CTCAE version 4.03, in combination with ascites and low albumin, in the absence of disease progression

SECONDARY OUTCOMES:
Tumor response based on radiologic assessment of MRI scans using mRECIST | Up to 6 months
  Tumor response based on radiologic assessment of MRI scans using mRECIST
Changes in tumor marker alpha-fetoprotein | Up to 6 months
  Changes in tumor marker alpha-fetoprotein
Quality of Life (QoL) using EORTC C30 | Up to 6 months
  Quality of Life (QoL) using EORTC C30
Quality of Life (QoL) using EORTC HCC18 | Up to 6 months
  Quality of Life (QoL) using EORTC HCC18
Quality of Life (QoL) using BPI-SF | Up to 6 months
  Quality of Life (QoL) using BPI-SF
Biodistribution/dosimetry based on quantitative assessment of MRI scans | Up to 6 months
  Biodistribution/dosimetry based on quantitative assessment of MRI scans
Changes in hepatic function as determined by hepatobiliary scintigraphy | Up to 3 months
  Changes in hepatic function as determined by hepatobiliary scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Marnix G. Lam, MD, PhD, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinders MTM, Smits MJL, van Erpecum K, de Bruijne J, Bruijnen RCG, Sprengers D, de Man R, Vegt E, IJzermans JNM, Lam MGEH, Braat AJAT. Hepatobiliary scintigraphy and liver function changes in patients with hepatocellular carcinoma treated with 166Ho-radioembolization : HBS in HCC treated with holmium-166. EJNMMI Res. 2025 Jan 9;15(1):2. doi: 10.1186/s13550-025-01196-9. PMID 39786516